CLINICAL TRIAL: NCT00443092
Title: A Double Blind Cross-over Study of the Efficacy of a Proprietary Cherry Juice Blend in Osteoarthritis of the Knee.
Brief Title: Efficacy of Proprietary Cherry Juice Blend in Osteoarthritis of the Knee
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CherryPharm (Industry)
Responsible Party: Brian Ross, Cherry Pharm
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CP100M; VA MIRB ID # 00981
Record Dates: First submitted 2007-03-02; First posted 2007-03-05 (Estimated); Last update posted 2012-08-03 (Estimated); Status verified 2012-08

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis; gout; pain; uric acid; tart cherry; alternative medicine; knees
MeSH Terms: conditions — Osteoarthritis; Gout; Pain | interventions — Food

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): proprietary tart cherry juice blend (8 oz., BID)
  Interventions: Other: proprietary cherry juice blend (food)
- 2 (Placebo Comparator): control juice (color matched kool aid blend),(8 oz., BID)
  Interventions: Other: control juice (kool aid blend)

INTERVENTIONS:
Other: proprietary cherry juice blend (food) — 2 bottles per day for 6 weeks, 1 in the morning and 1 in the evening
  Arms: 1
Other: control juice (kool aid blend) — 2 bottles per day for 6 weeks, 1 in the morning and 1 in the evening
  Arms: 2

SUMMARY:
The primary purpose of this research study is to test the ability of a proprietary cherry juice blend to be helpful in the treatment of osteoarthritis (OA) of the knee.

DETAILED DESCRIPTION:
The primary objective is to determine if the proprietary tart cherry juice blend improves the pain and function in persons with knee osteoarthritis. A secondary objective is to ascertain if the blend lowers serum uric acid.

This is a prospective double blind, placebo controlled cross-over study.

The study will be performed in the Philadelphia VA Medical Center 1 South Rheumatology Clinic with patients meeting ACR criteria for Kellgren grade 2-3 knee osteoarthritis and 4-9 pain severity on a VAS. Fifty patients will be studied with each having 5 visits. Subjects will take either the proprietary cherry blend or placebo for 6 weeks and then switch. WOMAC pain and function will be the primary outcome with acetaminophen use, walking time and serum uric acid as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Subject is capable of giving informed consent.
* Subject is over 18 years and less than 80 years
* Subject has mild to moderate osteoarthritis of the knee based on all of the following 3:

  1. Meets clinical ACR criteria
  2. Kellgren score of 2-3 on a Standing Knee x-ray within previous 24 months
  3. VAS pain score of 4-9 at screening visit

Exclusion Criteria:

* Rheumatoid arthritis or other systemic inflammatory condition
* Chronic pain syndrome (fibromyalgia)
* Corticosteroid medication in last 2 months, either intra-articular or oral
* Intra-articular injections of hyaluronic acid in last 9 months
* Pregnant women (weight gain might confound degree of knee pain)
* Diabetes
* Inability to discontinue prescription medication for arthritis
* Unstable medical conditions that would likely prevent the subject from completing the study
* Food allergies - cherries, apples

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2007-03; Primary Completion 2010-06 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Improvement in Western Ontario McMaster Osteoarthritis Index (WOMAC) Scores to be taken at Visits 2-5. | Visit 3 (week 6-7), Visit 5 (week 13-14)

SECONDARY OUTCOMES:
Determine if there is a decrease in amount of non-prescription pain medication taken and/or improvement in score on a timed walking test (Visits 2,3,4,5). | Visit 3 (week 6-7), Visit 5 (week 13-14)
Determine if there is a decrease in serum uric acid levels. (Visits 1,3,5) | Visit 3 (week 6-7), Visit 5 (week 13-14)

CONTACTS AND LOCATIONS:
Overall Officials: H. R Schumacher, M.D., Principal Investigator — VA Medical Center, Philadelphia & University of Pennsylvania
Locations (1):
- VA Medical Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] BLAU LW. Cherry diet control for gout and arthritis. Tex Rep Biol Med. 1950;8(3):309-11. No abstract available. PMID 14776685
- [Background] Connolly DA, McHugh MP, Padilla-Zakour OI, Carlson L, Sayers SP. Efficacy of a tart cherry juice blend in preventing the symptoms of muscle damage. Br J Sports Med. 2006 Aug;40(8):679-83; discussion 683. doi: 10.1136/bjsm.2005.025429. Epub 2006 Jun 21. PMID 16790484
- [Background] Seeram NP, Momin RA, Nair MG, Bourquin LD. Cyclooxygenase inhibitory and antioxidant cyanidin glycosides in cherries and berries. Phytomedicine. 2001 Sep;8(5):362-9. doi: 10.1078/0944-7113-00053. PMID 11695879
- [Background] He YH, Zhou J, Wang YS, Xiao C, Tong Y, Tang JC, Chan AS, Lu AP. Anti-inflammatory and anti-oxidative effects of cherries on Freund's adjuvant-induced arthritis in rats. Scand J Rheumatol. 2006 Sep-Oct;35(5):356-8. doi: 10.1080/03009740600704155. PMID 17062434
- [Background] Jacob RA, Spinozzi GM, Simon VA, Kelley DS, Prior RL, Hess-Pierce B, Kader AA. Consumption of cherries lowers plasma urate in healthy women. J Nutr. 2003 Jun;133(6):1826-9. doi: 10.1093/jn/133.6.1826. PMID 12771324
- [Background] Pincus T, Koch G, Lei H, Mangal B, Sokka T, Moskowitz R, Wolfe F, Gibofsky A, Simon L, Zlotnick S, Fort JG. Patient Preference for Placebo, Acetaminophen (paracetamol) or Celecoxib Efficacy Studies (PACES): two randomised, double blind, placebo controlled, crossover clinical trials in patients with knee or hip osteoarthritis. Ann Rheum Dis. 2004 Aug;63(8):931-9. doi: 10.1136/ard.2003.020313. Epub 2004 Apr 13. PMID 15082468
- [Background] Johanson NA, Liang MH, Daltroy L, Rudicel S, Richmond J. American Academy of Orthopaedic Surgeons lower limb outcomes assessment instruments. Reliability, validity, and sensitivity to change. J Bone Joint Surg Am. 2004 May;86(5):902-9. doi: 10.2106/00004623-200405000-00003. PMID 15118030
- [Background] Altman R, Asch E, Bloch D, Bole G, Borenstein D, Brandt K, Christy W, Cooke TD, Greenwald R, Hochberg M, et al. Development of criteria for the classification and reporting of osteoarthritis. Classification of osteoarthritis of the knee. Diagnostic and Therapeutic Criteria Committee of the American Rheumatism Association. Arthritis Rheum. 1986 Aug;29(8):1039-49. doi: 10.1002/art.1780290816. PMID 3741515